CLINICAL TRIAL: NCT02917070
Title: The Importance of Parental Consanguinity and Family History of Kidney Disease in Turkish Adult Chronic Kidney Disease Population
Brief Title: Parental Consanguinity and Family History of Kidney Disease in Turkish Kidney Disease Population
Acronym: CAKD
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Yasar Caliskan, Principal Investigator, Istanbul University
Other Study IDs: 2016/257; 301 (Registry Identifier: Yasar Calıskan)
Record Dates: First submitted 2016-09-09; First posted 2016-09-28 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-09

CONDITIONS: Hereditary Diseases
Keywords: Consanguinity-associated kidney diseases; Turkey population
MeSH Terms: conditions — Genetic Diseases, Inborn

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients: Patients who have chronic kidney diseases
  Interventions: Other: Patients
- Healthy controls: Healthy subjects

INTERVENTIONS:
Other: Patients — In this study we aimed to investigate effect of family history and consanguineous marriage in the development of CKD in the adult Turkish population.
  Other Names: Inbreeding marriage
  Groups: Patients

SUMMARY:
Inbreeding and consanguineous marriages are known to increase the risk of autosomal recessive disorders. The aim of this study was to examine the association between consanguinity and kidney diseases in the adult Turkish population.

DETAILED DESCRIPTION:
This was a national, cross-sectional study recruiting patients from nephrology out-patient clinics and dialysis units. All patients between 18 and 70 years of age who were on follow up in outpatient clinic and dialysis unit at the Istanbul Medical Faculty from October 2009 to October 2015 were included in the study. All patients and healthy controls enrolled in this study gave informed consent to participate in the survey. They were all asked to answer a questionnaire including socio-demographic data, history of familial kidney disease and consanguineous marriage. Additional information was obtained from their private physicians and medical files. To ensure reliability of administration of the questionnaire, all interviewers underwent training using a standardized protocol.

ELIGIBILITY:
Inclusion Criteria:

* follow up in outpatient clinic and dialysis unit at the Istanbul Medical Faculty
* between 18-70 years old
* provide informed consent

Exclusion Criteria:

* follow-up shorter than 6 months
* patients whose data were not available
* patients who were unwilling or unable to provide informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients between 18 and 70 years of age who were on follow up in outpatient clinic and dialysis unit at the Istanbul Medical Faculty from October 2009 to October 2015 were included in the study
Sampling Method: Non-Probability Sample
Enrollment: 2576 (Actual)
Dates: Start 2016-02; Primary Completion 2016-05 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Effect of parental consanguinity on chronic kidney disease confirmed by a questionnaire did they have consanguinity marriage or not. | 6 months after enrollment

SECONDARY OUTCOMES:
Effect of family history of kidney disease on the development of chronic kidney confirmed by a questionnaire did they have any parents with chronic kidney diseases or not. | 6 months after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Yasar Caliskan, Dr., Principal Investigator — Istanbul University, Istanbul Faculty of Medicine, Department of Internal Medicine, Division of Nephrology
Locations (1):
- Istanbul University, Istanbul Faculty of Medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] National Kidney Foundation. K/DOQI clinical practice guidelines for chronic kidney disease: evaluation, classification, and stratification. Am J Kidney Dis. 2002 Feb;39(2 Suppl 1):S1-266. No abstract available. PMID 11904577
- [Result] Chronic Kidney Disease Prognosis Consortium; Matsushita K, van der Velde M, Astor BC, Woodward M, Levey AS, de Jong PE, Coresh J, Gansevoort RT. Association of estimated glomerular filtration rate and albuminuria with all-cause and cardiovascular mortality in general population cohorts: a collaborative meta-analysis. Lancet. 2010 Jun 12;375(9731):2073-81. doi: 10.1016/S0140-6736(10)60674-5. Epub 2010 May 17. PMID 20483451
- [Result] Suleymanlar G, Utas C, Arinsoy T, Ates K, Altun B, Altiparmak MR, Ecder T, Yilmaz ME, Camsari T, Basci A, Odabas AR, Serdengecti K. A population-based survey of Chronic REnal Disease In Turkey--the CREDIT study. Nephrol Dial Transplant. 2011 Jun;26(6):1862-71. doi: 10.1093/ndt/gfq656. Epub 2010 Nov 4. PMID 21051501
- [Result] Gumprecht J, Zychma MJ, Grzeszczak W, Zukowska-Szczechowska E; End-stage Renal Disease Study Group. Human SA gene Pst1 polymorphism and chronic renal failure: results of the family-based study. Nephrol Dial Transplant. 2001 Feb;16(2):387-90. doi: 10.1093/ndt/16.2.387. PMID 11158418
- [Result] O'Dea DF, Murphy SW, Hefferton D, Parfrey PS. Higher risk for renal failure in first-degree relatives of white patients with end-stage renal disease: a population-based study. Am J Kidney Dis. 1998 Nov;32(5):794-801. doi: 10.1016/s0272-6386(98)70135-0. PMID 9820449